CLINICAL TRIAL: NCT06226727
Title: A Randomized, Open-label, Single Dose, Two-way Replicate Crossover Phase 1 Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR1019" and Co-administration of "BR1019-1" and "BR1019-2" in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and the Safety After Administration of "BR1019" and Co-administration of "BR1019-1" and "BR1019-2"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FDC-CT-103
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus; Essential Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence Group A (Experimental): The investigational products will be administered according to the treatment groups assigned to each sequence group in Period 1~4.
  *Sequence Group A [Period 1, 3] Co-administration of BR1019-1(R1) and BR1019-2(R2). [Period 2, 4] Administration of BR1019(T)
  Interventions: Drug: BR1019; Drug: BR1019-1; Drug: BR1019-2
- Sequence Group B (Experimental): The investigational products will be administered according to the treatment groups assigned to each sequence group in Period 1~4.
  *Sequence Group B [Period 1, 3] Administration of BR1019(T) [Period 2, 4] Co-administration of BR1019-1(R1) and BR1019-2(R2).
  Interventions: Drug: BR1019; Drug: BR1019-1; Drug: BR1019-2

INTERVENTIONS:
Drug: BR1019 — One tablet administered alone
Drug: BR1019-1 — One tablet administered alone
Drug: BR1019-2 — One tablet administered alone

SUMMARY:
The objective of this clinical study is to evaluate the pharmacokinetics and the safety after administration of "BR1019" and co-administration of "BR1019-1" and "BR1019-2" in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Those who have body mass index (BMI) within the range of 18.0 to 30.0kg/m² at screening visit

  * In case of a male subject, Those who weigh 50 kg or more
  * In case of a female subject, Those who weigh 45 kg or more
* Those who decide to voluntarily participate after listening to and understanding the detailed explanation of this clinical trial and who sign a written consent to comply with the subject's precautions during this clinical trial.

Exclusion Criteria:

* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 30 days prior to the first day of administration or have taken ETC, OTC, Oriental medicine, Health functional food concerned about affecting this clinical trial within 10 days prior to the first day of administration. (however, participation is possible considering pharmacokinetics and pharmacodynamics such as Interaction of investigational products, half-life of concomitant drugs, etc.)
* Those who have participated in bioequivalence tests or other clinical trials administered their investigational products within 6 months prior to the first administration date. (However, the termination for participation in other clinical trials are based on the last administration date of their investigational products)
* Those who have a medical history of gastrectomy(Except for simple appendectomy, hernia surgery) or gastrointestinal diseases that may affect the absorption of drugs.
* Those who can't discontinue a diet (ex. raw grapefruit, grapefruit juice or its products, etc.) that may affect the absorption, distribution, metabolism, and excretion of the drug within 48 hours prior to the first day of administration.
* In the case of a female subject, those suspected pregnancy, pregnant woman, lactating woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
AUCτ | 0-48 hours after administration
  Area under the concentration-time curve from time zero to time τ
Cmax | 0-48 hours after administration
  Maximum concentration of drug in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, Gwanakgu, South Korea

IPD SHARING:
Plan to Share IPD: No